CLINICAL TRIAL: NCT00288626
Title: A Phase II Study of High-Dose Immunosuppressive Therapy Using Carmustine, Etoposide, Cytarabine, Melphalan, Thymoglobulin and Autologous CD34+ Hematopoietic Stem Cell Transplant for the Treatment of Poor Prognosis Multiple Sclerosis
Brief Title: High-Dose Immunosuppression and Autologous Transplantation for Multiple Sclerosis (HALT MS) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN033AI; DAIT SCMS2
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: hematopoietic stem cell transplantation; HCT- autologous hematopoietic cell transplant; HDIT-high-dose immunosuppressive therapy; BEAM -Carmustine (BCNU), Etoposide (VP-16), Cytarabine (ara-C), and Melphalan
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Granulocyte Colony-Stimulating Factor; Prednisone; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MS Treatment (Experimental): Autologous peripheral blood stem cell grafts were CD34+ selected; the participants then received high-dose treatment with carmustine, etoposide, cytarabine, and melphalan as well as rabbit antithymocyte globulin before autologous HCT.
  Interventions: Drug: Granulocyte-colony stimulating factor (G-CSF) and prednisone; Drug: Carmustine, etoposide, cytarabine, and melphalan (BEAM); Procedure: Autologous hematopoietic stem cell transplant

INTERVENTIONS:
Drug: Granulocyte-colony stimulating factor (G-CSF) and prednisone — Growth factor regimen; occurs at study entry
Drug: Carmustine, etoposide, cytarabine, and melphalan (BEAM) — High-dose chemotherapy; occurs seven or more days following collection of autologous graft
Procedure: Autologous hematopoietic stem cell transplant — Occurs after growth factor regimen and collection of autologous graft

SUMMARY:
The purpose of this study is to determine the effectiveness of a new treatment for multiple sclerosis (MS), a serious disease in which the immune system attacks the brain and spinal cord. MS can be progressive and severe and lead to significant disability. The study treatment involves the use of high-dose chemotherapeutic drugs to suppress the immune system. The participant's own (autologous) blood-forming (hematopoietic, CD34+) stem cells are collected before the chemotherapy is given, and then transplanted back into the body following treatment. Transplantation of autologous hematopoietic stem cells is required to prevent very prolonged periods of low blood cell counts after the high-dose chemotherapy.

DETAILED DESCRIPTION:
MS is a chronic autoimmune disease of the central nervous system in which myelin, the protective coat that surrounds nerve cells, is damaged or destroyed by autoimmune T cells and macrophages, leading to an eventual loss of neurologic function. In a pilot study in Europe using high-dose chemotherapy, it was observed that 18 of 19 MS patients stabilized or improved clinically, and only one patient showed a new lesion on magnetic resonance imaging (MRI) of the brain at 4.5 years after treatment. Improvement was seen in quality-of-life assessments.

In ITN033AI, high-dose chemotherapy with autologous CD34-selected hematopoietic cell transplantation will be given to confirm the results from the pilot study and to offer therapy to patients with early MS and a poor prognosis. Research studies will be performed in addition to clinical assessments to better understand the effect of the treatment on the activity of MS. High-dose chemotherapy will be used to deplete autoreactive immune cells. These regimens also deplete the bone marrow, the source of blood-forming CD34+ stem cells which causes very low blood counts. Therefore, the participant's autologous CD34+ hematopoietic stem cells will be collected before high dose immunosuppressive therapy is given and then returned as a transplant post-chemotherapy. Patients will be followed closely after the autologous transplantation since they will be at risk for infections after treatment.

At the beginning of the study, participants will undergo a number of screening and baseline procedures, including a physical exam, blood collection, MS-confirming neurology exams and questionnaires, and MRI procedures. Participants will be given prednisone and granulocyte-colony stimulating factor (G-CSF) to mobilize CD34+ hematopoietic stem cells from the bone marrow into the peripheral blood. When the peripheral blood CD34+ cell count reaches 20,000 cells/ml or greater, these cells will be collected by leukapheresis. In this process, a catheter is placed into a large blood vessel, peripheral blood is withdrawn, and a high speed sedimentation (leukapheresis) device is used to separate and retain the cells required for autologous transplantation. Other blood cells are then returned to the participant's body. In the laboratory, the CD34+ hematopoietic stem cell graft will be selected and prepared from the leukapheresis collection, and stored until needed for transplant. Seven or more days following the collection of their autologous graft, participants will be hospitalized and receive high-dose chemotherapy consisting of carmustine, etoposide, cytarabine, and melphalan (BEAM) and thymoglobulin. This is followed by transplantation of the autologous hematopoietic cell graft. Participants will remain in the hospital for observation during recovery of their peripheral blood cell counts, as described in the protocol. Participants will receive G-CSF and blood transfusions, if needed, and will be monitored for infections. Following discharge from the hospital, eight study visits will occur over sixty months (five years). During these visits, participants will undergo blood and urine collection, MRI studies, leukapheresis, and MS neurology exams and will complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting or progressive-relapsing multiple sclerosis for less than 15 years using McDonald Criteria. More information on this criterion can be found in the protocol
* Score between 3.0 and 5.5 on the Expanded Disability Status Scale (EDSS)
* T2 abnormalities on brain MRI consistent with MS
* Two or more relapses in 18 months time on interferon (IFN), glatiramer acetate (GA), natalizumab or cytotoxic therapy with EDSS increase of 1.0 or greater for participants with EDSS at screening of 3.0 to 3.5 (0.5 or greater for participants with EDSS at screening of 4.0 to 5.5) sustained at least 4 weeks after at least one of these relapses OR one relapse on IFN, GA, natalizumab or cytotoxic therapy with EDSS increase of 1.5 or greater (1.0 for subjects with EDSS at screening of 5.5) sustained at least 4 weeks, together with MRI changes consistent with poor prognosis. More information on this criterion can be found in the protocol.
* On IFN or GA for at least 6 months before the relapses occur that are counted to satisfy previous inclusion criterion OR have received adequate doses of natalizumab or cytotoxic therapy on a treatment schedule before the relapses occur that are counted to satisfy previous inclusion criterion
* Approval by an MS Review Panel to participate in the study. More information on this criterion can be found in the protocol
* In good clinical condition with adequate organ function and without coexisting medical problems that would increase the risk to the participant
* Willing to use acceptable methods of contraception
* Willing and able to comply with all study requirements and
* Willing to accept and comprehend irreversible sterility as side effect of therapy.

Exclusion Criteria:

* Primary progressive MS
* Secondary progressive MS without relapses (i.e., progression without exacerbations or relapses) for 12 or more months
* Neuromyelitis optica, a disease similar to MS
* Initiation of new immunosuppressant treatment after the participant becomes eligible for the protocol or continuance of immunosuppressant drugs after the participant is screened for the protocol. Treatment with IFN, GA, or corticosteroids is permitted after the participant becomes eligible for the protocol.
* Lapse of greater than 6 months between the time a participant is eligible for the protocol and initiation of protocol treatment except when judged acceptable by the MS Review Panel
* Prior treatment with investigational immunosuppressive agents within 3 months of study eligibility
* Positive baseline plasma and CSF testing for JC virus or a brain MRI that has changes consistent with a diagnosis of progressive multifocal encephalopathy (PML)
* History of cytopenia consistent with the diagnosis of myelodysplastic syndrome (MDS)
* Active hepatitis B or C infection, cirrhosis, or HIV infection
* Uncontrolled diabetes mellitus
* Uncontrolled viral, fungal, or bacterial infection. Patients with asymptomatic bacteriuria are not excluded
* Any illness that would jeopardize the ability to tolerate aggressive chemotherapy
* Prior history of malignancy, except localized basal cell or squamous skin cancer. Other malignancies for which the subject is judged cured by the administered therapy will be considered on an individual basis.
* Hypersensitivity to mouse, rabbit, or Escherichia coli-derived proteins or to iron compounds/medications
* Metallic objects implanted in the body that would affect MRI exams
* Psychiatric illness, mental deficiency, or cognitive dysfunction or
* Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Nash, MD, Study Chair — Blood and Marrow Transplant Program, Colorado Blood Cancer Institute, Presbyterian/St. Luke's Medical Center, Denver; James D. Bowen, MD, Study Chair — Multiple Sclerosis Center, Swedish Neuroscience Institute, Seattle, Washington; George H. Kraft, MD, Study Chair — Departments of Neurology and Rehabilitation Medicine, University of Washington; George J. Hutton, MD, Study Chair — The Maxine Messinger Multiple Sclerosis Clinic, The Methodist Hospital, Baylor College of Medicine; Uday Popat, MD, Study Chair — Department of Blood and Marrow Transplantation, University of Texas, M.D. Anderson Cancer Center; Michael K. Racke, MD, Study Chair — Department of Neurology, Ohio State University Medical Center; Steven M. Devine, MD, Study Chair — Department of Hematology and Oncology, Ohio State University Medical Center; Annette Wundes, MD, Study Chair — Department of Neurology, University of Washington; George E. Georges, MD, Study Chair — Fred Hutchinson Cancer Research Center, Clinical Research Division, University of Washington
Locations (4):
- United States (4):
  - Ohio State University School of Medicine, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - M.D. Anderson Cancer Center; Transplant site, please contact Baylor College of Medicine, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data access is provided to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts that also provides data analysis tools available to researchers.

REFERENCES:
- [Background] Fassas A, Nash R. Stem cell transplantation for autoimmune disorders. Multiple sclerosis. Best Pract Res Clin Haematol. 2004 Jun;17(2):247-62. doi: 10.1016/j.beha.2004.04.005. PMID 15302338
- [Background] Muraro PA, Douek DC. Renewing the T cell repertoire to arrest autoimmune aggression. Trends Immunol. 2006 Feb;27(2):61-7. doi: 10.1016/j.it.2005.12.003. Epub 2006 Jan 6. PMID 16406806
- [Background] Muraro PA, Douek DC, Packer A, Chung K, Guenaga FJ, Cassiani-Ingoni R, Campbell C, Memon S, Nagle JW, Hakim FT, Gress RE, McFarland HF, Burt RK, Martin R. Thymic output generates a new and diverse TCR repertoire after autologous stem cell transplantation in multiple sclerosis patients. J Exp Med. 2005 Mar 7;201(5):805-16. doi: 10.1084/jem.20041679. Epub 2005 Feb 28. PMID 15738052
- [Background] Saccardi R, Mancardi GL, Solari A, Bosi A, Bruzzi P, Di Bartolomeo P, Donelli A, Filippi M, Guerrasio A, Gualandi F, La Nasa G, Murialdo A, Pagliai F, Papineschi F, Scappini B, Marmont AM. Autologous HSCT for severe progressive multiple sclerosis in a multicenter trial: impact on disease activity and quality of life. Blood. 2005 Mar 15;105(6):2601-7. doi: 10.1182/blood-2004-08-3205. Epub 2004 Nov 16. PMID 15546956
- [Background] Tyndall A, Saccardi R. Haematopoietic stem cell transplantation in the treatment of severe autoimmune disease: results from phase I/II studies, prospective randomized trials and future directions. Clin Exp Immunol. 2005 Jul;141(1):1-9. doi: 10.1111/j.1365-2249.2005.02806.x. PMID 15958063
- [Background] Mancardi G, Saccardi R. Autologous haematopoietic stem-cell transplantation in multiple sclerosis. Lancet Neurol. 2008 Jul;7(7):626-36. doi: 10.1016/S1474-4422(08)70138-8. PMID 18565456
- [Result] Nash RA, Hutton GJ, Racke MK, Popat U, Devine SM, Griffith LM, Muraro PA, Openshaw H, Sayre PH, Stuve O, Arnold DL, Spychala ME, McConville KC, Harris KM, Phippard D, Georges GE, Wundes A, Kraft GH, Bowen JD. High-dose immunosuppressive therapy and autologous hematopoietic cell transplantation for relapsing-remitting multiple sclerosis (HALT-MS): a 3-year interim report. JAMA Neurol. 2015 Feb;72(2):159-69. doi: 10.1001/jamaneurol.2014.3780. PMID 25546364
- [Result] Muraro PA, Robins H, Malhotra S, Howell M, Phippard D, Desmarais C, de Paula Alves Sousa A, Griffith LM, Lim N, Nash RA, Turka LA. T cell repertoire following autologous stem cell transplantation for multiple sclerosis. J Clin Invest. 2014 Mar;124(3):1168-72. doi: 10.1172/JCI71691. Epub 2014 Feb 17. PMID 24531550
- [Result] Nash RA, Hutton GJ, Racke MK, Popat U, Devine SM, Steinmiller KC, Griffith LM, Muraro PA, Openshaw H, Sayre PH, Stuve O, Arnold DL, Wener MH, Georges GE, Wundes A, Kraft GH, Bowen JD. High-dose immunosuppressive therapy and autologous HCT for relapsing-remitting MS. Neurology. 2017 Feb 28;88(9):842-852. doi: 10.1212/WNL.0000000000003660. Epub 2017 Feb 1. PMID 28148635
- [Result] Keever-Taylor CA, Heimfeld S, Steinmiller KC, Nash RA, Sullivan KM, Czarniecki CW, Granderson TC, Goldstein JS, Griffith LM. Manufacture of Autologous CD34+ Selected Grafts in the NIAID-Sponsored HALT-MS and SCOT Multicenter Clinical Trials for Autoimmune Diseases. Biol Blood Marrow Transplant. 2017 Sep;23(9):1463-1472. doi: 10.1016/j.bbmt.2017.05.018. Epub 2017 Jun 30. PMID 28602891
- [Derived] Harris KM, Lu T, Lim N, Turka LA. Challenges and Opportunities for Biomarkers of Clinical Response to AHSCT in Autoimmunity. Front Immunol. 2018 Feb 2;9:100. doi: 10.3389/fimmu.2018.00100. eCollection 2018. PMID 29456529
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY549 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY549 — Deidentified participant ID mapping to manuscript ID. ImmPort study identifier is SDY549.
- Available data/document: Study summary, -design, -demographics, and -study files — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY549 — ImmPort study identifier is SDY549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 participants were screened and 25 of those participants were enrolled at 3 sites in the US between August 2006 and August 2009. 24 participants were transplanted with the cellular product between February 2007 and April 2010
Groups:
- HDIT and HCT: Participants recv'd Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until ≥ 2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to > 500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Period: Overall Study
Arm/Group | HDIT and HCT
Started | 24
Completed | 17
Not Completed | 7
Not completed — Death | 3
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Participants who received High-Dose Immunosuppressive Therapy (HDIT)and Autologous CD34+ Hematopoietic Stem Cell Transplant (HCT)
Groups:
- HDIT and HCT: Participants recv'd Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until ≥2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to > 500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Expanded Disability Status Scale (EDSS) at Baseline [Mean (Standard Deviation); unit: units on a scale] — Kurtzke's Expanded Disability Status Scale (EDSS) assesses disability in Multiple Sclerosis patients. Eight functional systems are evaluated: visual, brain stem, pyramidal, cerebellar, sensory, bowel and bladder, cerebral, and ambulation. The overall score ranges from 0 (normal neurological exam) to 10 (death due to MS).
  units on a scale | 4.4 (.64)
Number of Gadolinium-Enhanced Lesions at Baseline [Mean (Standard Deviation); unit: Lesions per scan] — Multiple sclerosis disease-related lesions were assessed by gadolinium-enhanced magnetic resonance imaging (MRI). More lesions indicate more severe disease.
  Lesions per scan | 2.3 (5.8)
T1 Lesion Volume at Baseline [Mean (Standard Deviation); unit: milliliters] — A T1-weighted magnetic resonance imaging (MRI) scan assessed the volume of T1 lesions.
  milliliters | 1.2 (2.7)
T2 Lesion Volume at Baseline [Mean (Standard Deviation); unit: milliliters] — A T2-weighted magnetic resonance imaging (MRI) scan assessed the volume of T2 lesions in the brain.
  milliliters | 11.1 (13.7)
Normalized Brain Volume at Screening [Mean (Standard Deviation); unit: liters] — Magnetic resonance imaging (MRI) scan techniques measured ventricular volumes and grey and white matter brain volumes
  liters | 1.6 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival Probability During the 5 Years After Transplant
Description: Event-free survival (EFS) is survival without death or disease activity from any one of the following criteria: 1) loss of neurological function, defined as a change in pretransplant Extended Disability Status Scale (EDSS) of > 0.5. 2) Relapse, defined as the development of a new neurological sign and corresponding symptom, or worsening of an existing neurological sign and symptom, localized to central nervous system white matter, resulting in neurological deficit/disability, and lasting over 48 hours. 3) New lesions on magnetic resonance imaging (MRI), defined as presence of 2 or more independent multiple sclerosis brain lesions detected on MRI 1 year or more after stem cell transplant. Kaplan-Meier estimates of survival probability, with 90% confidence interval based on Greenwood's formula for standard error.
Time Frame: 5 years
Population: Participants who received High-Dose Immunosuppressive Therapy (HDIT) and Autologous CD34+ Hematopoietic Stem Cell Transplant (HCT).
Measure: Number (90% Confidence Interval); unit: Probability
Groups:
- HDIT and HCT: Participants recv'd Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until ≥2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to >500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability | 0.692 [0.502 to 0.821]

2. Secondary Outcome: Event-Free Survival Probability During the 3 Years After Transplant
Description: as for outcome 1
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Groups:
- HDIT and HCT: Participants received Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until ≥2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to > 500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability | 0.784 [0.601 to 0.890]

3. Secondary Outcome: Survival From Treatment-Related Mortality
Description: The probability that a participant did not experienced a treatment-related death estimated at 1, 2, 3, 4, and 5 years following transplant via the Kaplan-Meier Method. Greenwood's formula for standard error was used to calculate 90% confidence intervals. Participants that did not experience a treatment-related death were censored at the time of last follow-up. A treatment-related death was defined as death that occurred at any time after study entry and that was possibly, probably, or definitely related to the cellular product or possibly, probably, or definitely related to mobilization of autologous peripheral blood hematopoietic progenitor cells with G-CSF and prednisone or to the high-dose immunosuppressive therapy. There were no treatment-related mortality events in the study.
Time Frame: From study entry to death, loss to follow-up, or the end of the study, whichever came first, up to 6 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Groups:
- HDIT and HCT: Participants recv'd Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until ≥ 2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to >500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 1.0 [1.0 to 1.0]
  2 Years Post Transplant | 1.0 [1.0 to 1.0]
  3 Years Post Transplant | 1.0 [1.0 to 1.0]
  4 Years Post Transplant | 1.0 [1.0 to 1.0]
  5 Years Post Transplant | 1.0 [1.0 to 1.0]

4. Secondary Outcome: Overall Survival
Description: The probability that a participant did not experienced a death estimated at 1, 2, 3, 4, and 5 years following transplant via the Kaplan-Meier Method. Greenwood's formula for standard error was used to calculate 90% confidence intervals. Participants that did not die were censored at the time of last follow-up.
Time Frame: From study entry to death, loss to follow-up, or the end of the study, whichever came first, up to 6 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 1.0 [1.0 to 1.0]
  2 Years Post Transplant | 1.0 [1.0 to 1.0]
  3 Years Post Transplant | 0.957 [0.794 to 0.991]
  4 Years Post Transplant | 0.911 [0.742 to 0.971]
  5 Years Post Transplant | 0.863 [0.683 to 0.945]

5. Secondary Outcome: Survival From MS-Related Mortality
Description: The probability that a participant did not experienced a MS-related death estimated at 1, 2, 3, 4, and 5 years following transplant via the Kaplan-Meier Method. Greenwood's formula for standard error was used to calculate 90% confidence intervals. Participants that did not experience a MS-related death were censored at the time of last follow-up. A MS-related death was defined as death that occurred at any time after study entry and that was possibly, probably, or definitely related to disease progression.
Time Frame: From study entry to death, loss to follow-up, or the end of the study, whichever came first, up to 6 years
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 1.0 [1.0 to 1.0]
  2 Years Post Transplant | 1.0 [1.0 to 1.0]
  3 Years Post Transplant | 0.957 [0.794 to 0.991]
  4 Years Post Transplant | 0.957 [0.794 to 0.991]
  5 Years Post Transplant | 0.906 [0.728 to 0.970]

6. Secondary Outcome: Percent of Participants Who Experienced All-Cause Morbidity
Description: Morbidity is the occurrence of NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0 adverse event grade 3 or higher.
Time Frame: From the time of enrollment until completion of the 5-year follow-up, an average of 6 years.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
percentage of participants | 100

7. Secondary Outcome: Percent of Participants Who Experienced All-Cause Morbidity Within 12 Months of Post-HCT
Description: as for outcome 6
Time Frame: From the time of Autologous CD34+ Hematopoietic Stem Cell Transplant (HCT) to 1 year after HCT.
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Percentage of Participants | 95.8

8. Secondary Outcome: Time to Neutrophil Engraftment
Description: Neutrophil engraftment, or neutrophil count recovery, is defined as an Absolute Neutrophil Count (ANC) > 500/ μL for 2 consecutive measurements on different days. Normal range is 1500 to 8000/μL. Reference: http://www.medicinenet.com
Time Frame: From time of graft infusion to time of engraftment, up to 6 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Days | 10.8 (1.1)

9. Secondary Outcome: Time to Platelet Engraftment
Description: Platelet engraftment, or platelet count recovery, is defined as Platelets > 20,000/μL for two consecutive measurements on different days with no platelet transfusions in the preceding 7 days. Normal range is 150,000-450,000/μL. Reference: http://www.hopkinsmedicine.org/heart_vascular_institute/clinical_services/centers_excellence/womens_cardiovascular_health_center/patient_information/health_topics/platelets.html.
Time Frame: From time of graft infusion to time of engraftment, up to 6 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Days | 18.5 (3.4)

10. Secondary Outcome: Event-Free Survival Probability After Transplant
Description: Event-free survival (EFS) is survival without death or disease activity from any one of the following criteria: 1) loss of neurological function, defined as a change in pretransplant Extended Disability Status Scale (EDSS) of > 0.5. 2) Relapse, defined as the development of a new neurological sign and corresponding symptom, or worsening of an existing neurological sign and symptom, localized to central nervous system white matter, resulting in neurological deficit/disability, and lasting over 48 hours. 3) New lesions on magnetic resonance imaging (MRI), defined as presence of 2 or more independent multiple sclerosis brain lesions detected on MRI 1 year or more after stem cell transplant. Kaplan-Meier estimates of survival probability, with 90% confidence intervals based on Greenwood's formula for standard error.
Time Frame: 1, 2, and 4 years after HCT
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 0.958 [0.802 to 0.992]
  2 Years Post Transplant | 0.828 [0.650 to 0.920]
  4 Years Post Transplant | 0.738 [0.550 to 0.857]

11. Secondary Outcome: MS Progression-Free Survival Probability After Transplant
Description: MS progression is measured as number of days from transplant to first Kurtzke's Expanded Disability Status Scale (EDSS) increase of more than 0.5 relative to the baseline measurement. EDSS assesses disability in Multiple Sclerosis patients. Eight functional systems are evaluated: visual, brain stem, pyramidal, cerebellar, sensory, bowel and bladder, cerebral, and ambulation. The overall score ranges from 0 (normal neurological exam) to 10 (death due to MS).
  Kaplan-Meier estimates of survival probability, with 90% confidence intervals based on Greenwood's formula for standard error.
Time Frame: 1 to 5 years after HCT
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 1.0 [1.0 to 1.0]
  2 Years Post Transplant | 0.913 [0.747 to 0.972]
  3 Years Post Transplant | 0.913 [0.747 to 0.972]
  4 Years Post Transplant | 0.913 [0.747 to 0.972]
  5 Years Post Transplant | 0.913 [0.747 to 0.972]

12. Secondary Outcome: MRI Activity-Free Survival Probability After Transplant
Description: MS disease activity is measured as days from transplant to first occurrence of >= 2 new MS lesions on Magnetic resonance imaging (MRI) relative to baseline. Kaplan-Meier estimates of survival probability, with 90% confidence intervals based on Greenwood's formula for standard error.
Time Frame: 1 to 5 years after HCT
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 0.958 [0.802 to 0.992]
  2 Years Post Transplant | 0.958 [0.802 to 0.992]
  3 Years Post Transplant | 0.958 [0.802 to 0.992]
  4 Years Post Transplant | 0.910 [0.739 to 0.971]
  5 Years Post Transplant | 0.863 [0.681 to 0.945]

13. Secondary Outcome: MS Relapse-Free Survival Probability After Transplant
Description: MS clinical relapse is defined as the development of a new neurological sign and corresponding symptom, or worsening of an existing neurological sign and symptom, localized to central nervous system white matter, resulting in neurological deficit or disability, and lasting over 48 hours. Clinical relapse was determined by the participant's neurologist and was measured as days from transplant to new or worsening neurological symptom relative to baseline.
  Kaplan-Meier estimates of survival probability, with 90% confidence interval based on Greenwood's formula for standard error.
Time Frame: 1 to 5 years after HCT
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 0.958 [0.802 to 0.992]
  2 Years Post Transplant | 0.915 [0.752 to 0.973]
  3 Years Post Transplant | 0.869 [0.695 to 0.947]
  4 Years Post Transplant | 0.869 [0.695 to 0.947]
  5 Years Post Transplant | 0.869 [0.695 to 0.947]

14. Secondary Outcome: Disease-Modifying Therapy Survival Probability After Transplant
Description: Treatment with disease-modifying therapy was measured by the number of days from transplant to the first treatment with an additional disease-modifying therapy. Examples of therapy include interferon beta-1a, glatiramer acetate, natalizumab, alemtuzumab, other immunosuppressive medications, or experimental therapies directed against MS activity. Kaplan-Meier estimates of survival probability, with 90% confidence interval based on Greenwood's formula for standard error.
Time Frame: 1 to 5 years after HCT
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Probability
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Probability
  1 Year Post Transplant | 1.0 [1.0 to 1.0]
  2 Years Post Transplant | 1.0 [1.0 to 1.0]
  3 Years Post Transplant | 1.0 [1.0 to 1.0]
  4 Years Post Transplant | 1.0 [1.0 to 1.0]
  5 Years Post Transplant | 0.950 [0.767 to 0.990]

15. Secondary Outcome: Change From Baseline in Extended Disability Status Scale (EDSS)
Description: Kurtzke's Expanded Disability Status Scale (EDSS) assesses disability in Multiple Sclerosis patients. Eight functional systems are evaluated: visual, brain stem, pyramidal, cerebellar, sensory, bowel and bladder, cerebral, and ambulation. The overall score ranges from 0 (normal neurological exam) to 10 (death due to MS). Change from baseline was computed as the value at the time point minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening. A change of > 0.5 in EDSS was a treatment-failure criterion.
Time Frame: 6 months to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
units on a scale
  6 Months Post Transplant | -0.3 (1.0)
  1 Year Post Transplant | -0.7 (0.9)
  2 Years Post Transplant | -0.8 (1.1)
  3 Years Post Transplant | -0.8 (1.1)
  4 Years Post Transplant | -0.6 (1.2)
  5 Years Post Transplant | -0.9 (1.0)

16. Secondary Outcome: Change From Baseline in Number of Gadolinium-Enhanced Lesions
Description: Multiple sclerosis disease-related lesions were assessed by gadolinium-enhanced magnetic resonance imaging (MRI). Change from baseline was computed as the value at the time point minus the baseline value. A negative value in change from baseline indicates an improvement and a positive value indicates worsening.
Time Frame: 8 weeks to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesions per scan
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Lesions per scan
  8 Weeks Post Transplant | -2.1 (4.9)
  6 Months Post Transplant | -2.3 (6.0)
  1 Year Post Transplant | -2.5 (6.1)
  2 Years Post Transplant | -2.5 (6.1)
  3 Years Post Transplant | -1.3 (2.2)
  4 Years Post Transplant | -2.2 (6.7)
  5 Years Post Transplant | -2.7 (7.0)

17. Secondary Outcome: Number of New T2-Weighted Lesions From Baseline
Description: A T2-weighted magnetic resonance imaging (MRI) scan was used to determine the number of new T2 lesions in the brain relative to Baseline. A value of 0 means that the participant didn't worsen. Values greater than 0 indicate an increase in disease activity from baseline.
Time Frame: 6 Months to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Lesions per scan
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Lesions per scan
  6 Months Post Transplant | 0.2 (0.5)
  1 Year Post Transplant | 0.2 (0.5)
  2 Years Post Transplant | 0.2 (0.5)
  3 Years Post Transplant | 0.1 (0.3)
  4 Years Post Transplant | 0.4 (1.2)
  5 Years Post Transplant | 0.1 (0.3)

18. Secondary Outcome: Change From Baseline in T2-Weighted Lesion Volume
Description: A T2-weighted magnetic resonance imaging (MRI) scan was used to assess the volume of T2 lesions in the brain. Change from baseline was computed as the value at the time point minus the baseline value.
Time Frame: 8 weeks to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
milliliters
  8 Weeks Post Transplant | -0.8 (1.9)
  6 Months Post Transplant | -0.7 (1.5)
  1 Year Post Transplant | -1.0 (1.6)
  2 Years Post Transplant | -1.6 (3.0)
  3 Years Post Transplant | -1.9 (3.1)
  4 Years Post Transplant | -1.9 (3.2)
  5 Years Post Transplant | -2.3 (3.6)

19. Secondary Outcome: Change From Baseline in T1-Weighted Lesion Volume
Description: A T1-weighted magnetic resonance imaging (MRI) scan was used to assess the volume of T1 lesions in the brain. Change from baseline was computed as the value at the time point minus the baseline value.
Time Frame: 8 weeks to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
milliliter
  8 Weeks Post Transplant | -0.1 (0.4)
  6 Months Post Transplant | 0.0 (0.4)
  1 Year Post Transplant | 0.2 (0.4)
  2 Years Post Transplant | 0.3 (0.7)
  3 Years Post Transplant | 0.4 (0.6)
  4 Years Post Transplant | 0.4 (0.7)
  5 Years Post Transplant | 0.3 (0.7)

20. Secondary Outcome: Percent Change From Screening in Brain Volume
Description: Magnetic resonance imaging (MRI) scan techniques measured ventricular volumes and grey and white matter brain volumes. Change from screening was computed as the value at the time point minus the screening value.
Time Frame: 8 weeks to 5 years after HCT
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | HDIT and HCT
Number analyzed (Participants) | 24
Percent Change
  8 Weeks Post Transplant | -0.8 (0.8)
  6 Months Post Transplant | -1.1 (0.9)
  1 Year Post Transplant | -1.2 (1.1)
  2 Years Post Transplant | -1.6 (1.4)
  3 Years Post Transplant | -2.2 (1.4)
  4 Years Post Transplant | -2.0 (1.4)
  5 Years Post Transplant | -2.3 (1.6)

ADVERSE EVENTS:
Time Frame: From the time the participant signed informed consent until the participant completed the 5-year follow-up, an average of 6 years
Description: Adverse events were reported for all participants enrolled. One participant in the group did not receive a transplant and was followed for safety only, no other analyses were performed for this participant.
Groups:
- HDIT and HCT: Participants recv'd Granulocyte Colony Stimulating Factor (G-CSF) by injection for 4-5 days to increase the number of blood stem cells in the blood stream by mobilizing them from the bone marrow. Leukapheresis was performed until > 2.0 x 10^6 CD34+ hematopoietic progenitor cells (HPCs) per kg were collected and frozen for future use. After ≥7 days following the last G-CSF dose, patients were hospitalized and received high-dose immunosuppression (HDIT) and immunosuppressive agent thymoglobulin 2.5 mg/kg over the course of 6 days. HDIT consisted of carmustine 300mg/m^2, etoposide 200 mg/m^2 cytarabine 200 mg/m^2, and melphalan 140 mg/m^2. CD34+ HPCs were thawed and infused according to institutional best practice for blood component transfusion over approximately 30 minutes. Patients were hospitalized until recovery of ANC to > 500/uL for at least 2 days. Prednisone was administered (0.5 mg/kg/day) from Days 7 to 21 after HCT and tapered over 2 weeks to prevent engraftment syndrome.
Arm/Group | HDIT and HCT
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDIT and HCT (N=25)
Leukopenia (Blood and lymphatic system disorders) | 2 (3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (4)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Engraftment syndrome (Immune system disorders) | 1 (1)
Acinetobacter infection (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2)
Motor dysfunction (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 3 (3)
Neurological symptom (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 1 (2)
Mania (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDIT and HCT (N=25)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 22 (31)
Lymphopenia (Blood and lymphatic system disorders) | 25 (48)
Neutropenia (Blood and lymphatic system disorders) | 23 (27)
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (25)
Hypothyroidism (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Gastritis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (10)
Chest pain (General disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 3 (5)
Bronchitis (Infections and infestations) | 2 (2)
Catheter site infection (Infections and infestations) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 6 (6)
Herpes zoster (Infections and infestations) | 7 (8)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 5 (9)
Urinary tract infection (Infections and infestations) | 7 (12)
Radius fracture (Injury, poisoning and procedural complications) | 2 (3)
Alanine aminotransferase increased (Investigations) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (6)
Multiple sclerosis (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Hypotension (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
24 of the 25 planned transplants occurred. One of the enrolled participants developed adverse events that caused withdrawal from the study before the planned transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No